CLINICAL TRIAL: NCT07055048
Title: The Diagnostic Efficacy and Lesion Detection Advantages of 18F-FDG PET/Contrast-enhanced MRI in Malignant Liver Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024YS-212
Record Dates: First submitted 2025-06-24; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer, Adult
Keywords: PET/MR; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research group: It is expected to include 60 patients with suspected hepatic space-occupying lesions , and the tracer radiation used in the study is extremely small and will not have any physiological effects on the subjects.

SUMMARY:
Liver disease, a major global health burden, ranges from mild dysfunction to severe conditions like cirrhosis and hepatocellular carcinoma (HCC), the fifth most common cancer. Accurate diagnosis of liver lesions-distinguishing benign from malignant-is vital for treatment planning. Conventional imaging (ultrasound, CT, MRI) has limitations in sensitivity and detecting small metastases. PET/CT combines metabolic and anatomical data but struggles with small lesions and cirrhotic livers.

18F-FDG PET/MRI with contrast-enhanced MRI may improve diagnostic accuracy, but its clinical benefits remain uncertain. Further research is needed to evaluate its performance, impact on patient outcomes, and cost-effectiveness in liver disease management.

DETAILED DESCRIPTION:
Liver disease is a major global public health challenge, ranging from mild dysfunction to severe conditions like cirrhosis and liver cancer. The high morbidity and mortality of liver diseases impose a significant socioeconomic burden, especially in developing countries. Primary liver cancer, particularly hepatocellular carcinoma (HCC), ranks as the fifth most common cancer and the third leading cause of cancer-related deaths worldwide. Additionally, the liver is a frequent site for metastases, and their presence critically impacts patient prognosis and treatment strategies.

Accurate diagnosis of liver lesions is essential for improving patient outcomes. Distinguishing benign from malignant lesions helps avoid unnecessary invasive procedures and ensures timely treatment. Similarly, early detection of liver metastases is crucial for cancer management and survival.

Conventional imaging techniques-such as ultrasound, CT, and MRI-are widely used for liver lesion assessment but have limitations, including insufficient specificity/sensitivity and difficulty in detecting small metastases. PET/CT, combining metabolic and anatomical data, is valuable in oncology but has drawbacks in liver applications, such as limited resolution for small lesions and challenges in differentiating malignancies in cirrhotic livers. Radiation exposure from CT is another concern.

In contrast, 18F-FDG PET/MRI with contrast-enhanced abdominal MRI offers a promising alternative, potentially improving diagnostic accuracy. However, despite its theoretical advantages, the actual clinical benefits remain unclear. A comprehensive study is needed to evaluate its diagnostic performance, accuracy, and impact on patient outcomes. Such research would validate its clinical utility, guide optimized treatment strategies, and ensure cost-effective integration into liver disease management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patients with suspected liver metastases or hepatic lesions,
* Ability to undergo 18F-FDG PET/MRI examination;
* Willingness to comply with study protocols.

Exclusion Criteria:

* Patients with a history of allergic reactions to MRI contrast agents;
* Pregnant or lactating women;
* Patients with severe comorbidities, including: Cardiac disease，Renal failure，or Hepatic failure (Child-Pugh C);
* Patients unable to cooperate with PET/MRI procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion and exclusion criteria and are willing to follow the research process.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic parameters | After the patient completes the scan, an average of 2 days.
  For all liver lesions, the maximum standardized uptake value (SUVmax) will be calculated.
MRI enhancement pattern | After the patient completes the scan, an average of 2 days.
  The MRI protocol will specifically evaluate the dynamic contrast-enhanced patterns of lesions, including their enhancement characteristics during the arterial phase, portal venous phase, and delayed phase.
Normal liver SUVmax | After the patient completes the scan, an average of 2 days.
  Calculate the maximum standardized uptake value (SUVmax) of normal liver tissue surrounding the lesion.

IPD SHARING:
Plan to Share IPD: No
For the protection of patient privacy, we will not share patient information, but other researchers can apply through the project contact person if they have reasonable reasons.